CLINICAL TRIAL: NCT02400814
Title: Pilot Study of MPDL3280A Plus Stereotactic Ablative Radiotherapy (SAR) in Stage IV Non-small Cell Lung Cancer
Brief Title: MPDL3280A and Stereotactic Ablative Radiotherapy in Patients With Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment halted due to slow accrual.
Sponsor: Megan Daly, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Megan Daly, MD, Professor of Clinical Radiation Oncology, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 685389; UCDCC#251 (CTRP (Clinical Trial Reporting Program)); ML29551; UCDCC#251 (Other: University of California, Davis); P30CA093373 (NIH); NCI-2014-02629 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-01-22; First posted 2015-03-27 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Recurrent Non-Small Cell Lung Carcinoma; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (concurrent cohort) (Experimental): Patients receive anti-PD-L1 monoclonal antibody MPDL3280A IV over 30-60 minutes on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Beginning on day 1 of course 1, patients also undergo SAR 2-3 times per week (with a minimum of 40 hours and a maximum of 96 hours between fractions) over 1.5-2 weeks for a total of 5 fractions.
  Interventions: Drug: Anti-PD-L1 Monoclonal Antibody MPDL3280A; Radiation: Stereotactic Body Radiation Therapy
- Arm II (induction cohort) (Experimental): Patients receive anti-PD-L1 monoclonal antibody MPDL3280A IV over 30-60 minutes on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Beginning on day 1 of course 3, patients also undergo SAR 2-3 times per week (with a minimum of 40 hours and a maximum of 96 hours between fractions) over 1.5-2 weeks for a total of 5 fractions.
  Interventions: Drug: Anti-PD-L1 Monoclonal Antibody MPDL3280A; Radiation: Stereotactic Body Radiation Therapy
- Arm III (sequential cohort) (Experimental): Patients undergo SAR 2-3 times per week (with a minimum of 40 hours and a maximum of 96 hours between fractions) over 1.5-2 weeks for a total of 5 fractions beginning on day 1 of course 1. After completion of SAR (beginning on day 1 of course 2), patients receive anti-PD-L1 monoclonal antibody MPDL3280A IV over 30-60 minutes on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Anti-PD-L1 Monoclonal Antibody MPDL3280A; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Anti-PD-L1 Monoclonal Antibody MPDL3280A — Given IV
  Other Names: MPDL3280A; RG7446
Radiation: Stereotactic Body Radiation Therapy — Undergo SAR
  Other Names: SBRT

SUMMARY:
This pilot phase I trial compares administration schedules of anti-programmed cell death-1 ligand 1 (PD-L1) monoclonal antibody MPDL3280A and stereotactic ablative radiotherapy in treating patients with stage IV non-small cell lung cancer. Monoclonal antibodies, such as anti-PD-L1 monoclonal antibody MPDL3280A, may block tumor growth in different ways by targeting certain cells. Stereotactic ablative radiotherapy, also known as stereotactic body radiation therapy, is a specialized radiation therapy that delivers a single, high dose of radiation directly to the tumor and may kill more tumor cells and cause less damage to normal tissue. Giving anti-PD-L1 monoclonal antibody MPDL3280A with stereotactic ablative radiotherapy may be a better treatment for non-small cell lung cancer. However, it is not yet known what the best administration schedule is for these treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine which administration schedule of MPDL3280A (anti-PD-L1 monoclonal antibody MPDL3280A) and stereotactic ablative radiotherapy (SAR) will be most promising to move forward to a phase II trial based on safety and objective response rate.

SECONDARY OBJECTIVES:

I. To define the safety and toxicity profile of MPDL3280A plus SAR using Common Terminology Criteria for Adverse Events (CTCAE) version 4 (v4).

II. Radiographic response rates by immure-related Response Evaluation Criteria in Solid Tumors (irRECIST).

III. Progression free survival using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and irRECIST.

TERTIARY OBJECTIVES:

I. Conduct correlative immunologic endpoints.

OUTLINE: Patients are assigned to 1 of 3 arms.

ARM I (CONCURRENT COHORT): Patients receive anti-PD-L1 monoclonal antibody MPDL3280A intravenously (IV) over 30-60 minutes on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Beginning on day 1 of course 1, patients also undergo SAR 2-3 times per week (with a minimum of 40 hours and a maximum of 96 hours between fractions) over 1.5-2 weeks for a total of 5 fractions.

ARM II (INDUCTION COHORT): Patients receive anti-PD-L1 monoclonal antibody MPDL3280A IV over 30-60 minutes on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Beginning on day 1 of course 3, patients also undergo SAR 2-3 times per week (with a minimum of 40 hours and a maximum of 96 hours between fractions) over 1.5-2 weeks for a total of 5 fractions.

ARM III (SEQUENTIAL COHORT): Patients undergo SAR 2-3 times per week (with a minimum of 40 hours and a maximum of 96 hours between fractions) over 1.5-2 weeks for a total of 5 fractions beginning on day 1 of course 1. After completion of SAR (beginning on day 1 of course 2), patients receive anti-PD-L1 monoclonal antibody MPDL3280A IV over 30-60 minutes on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Ability to comply with the protocol
* Adults with histologically proven stage IV non-small cell lung cancer
* At least two sites of measurable disease as defined by RECIST 1.1; one of which must be amenable to treatment with SAR and accessible for optional pre- and post- treatment biopsy; if a pulmonary nodule is being considered for SAR it must range in size from 1-3 cm
* Have provided written consent for mandatory pre- and post-treatment biopsy (expansion cohort only)
* Patients with treated supratentorial metastases are allowed if stable, the patient is off steroids and no evidence of intracranial hemorrhage
* Archival tumor sample available; a minimum of 10 unstained slides; no fine needle aspiration (FNAs) allowed or tumor tissue from bone
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Life expectancy >= 3 months
* Absolute neutrophil count (ANC) >= 1500 cells/ul
* White blood cell (WBC) count > 2500/uL
* Lymphocyte count >= 500/uL
* Platelet count >= 100,000/uL
* Hemoglobin >= 9 g/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x upper limit of normal (ULN) with alkaline phosphatase =< 2.5 x ULN OR AST and ALT =< 1.5 x ULN, with alkaline phosphatase > 2.5 x ULN
* Serum bilirubin =< 1.0 x ULN
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN (for patients on anticoagulation they must be receiving a stable dose for at least 1 week prior to randomization)
* Creatinine clearance >= 30 mL/min by Cockcroft-Gault formula
* No history of severe hypersensitivity reactions to other monoclonal antibodies (mAbs)
* No other active malignancy
* No active autoimmune disease or a history of known or suspected autoimmune disease
* No chemotherapy or radiotherapy within the past 28 days and patients must have recovered any acute toxicity associated with their most recent previous treatment
* Any number of prior treatments is allowed; must have failed at least 1 treatment regimen for metastatic disease
* Female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use highly effective form(s) of contraception

Exclusion Criteria:

* Patients whose tumors contain activating epidermal growth factor receptor (EGFR) mutations or anaplastic lymphoma receptor tyrosine kinase (ALK) rearrangement should be excluded from this study, unless disease has progressed on all available, approved therapies targeting the EGFR mutation or ALK rearrangement
* Active or untreated central nervous system (CNS) metastases
* Leptomeningeal disease
* Uncontrolled pleural or pericardial effusion or ascites that would require recurrent drainage
* Uncontrolled tumor related pain
* Uncontrolled hypercalcemia
* Pregnant and lactating women
* Uncontrolled concomitant disease
* Significant cardiovascular disease (New York Heart Association class II or greater); myocardial infarction within 3 months prior to enrollment, unstable arrhythmias, unstable angina or a patient with a known left ventricular ejection fraction (LVEF) < 40%
* Severe infection within 4 weeks prior to enrollment
* Oral or IV antibiotics within 2 weeks prior to enrollment
* History of severe allergic, anaphylactic or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity or allergy to Chinese hamster ovary cell products or any component of the MDPL3280A formulation
* History of autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis

  * Patients with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible
  * Patients with controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible
* Patients with a prior allogeneic bone marrow transplantation or prior solid organ transplantation
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e. bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest computed tomography (CT) scan

  * A history of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Positive test for human immunodeficiency virus (HIV)
* Patients with active hepatitis B (defined as a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C

  * Patients with past hepatitis B virus infection or resolved hepatitis B virus (HBV) infection (defined as a negative HBSAg test and a positive antibody to hepatitis B core antigen antibody test) are eligible
  * Patients with a hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA)
* Active tuberculosis
* Administration of a live, attenuated vaccine within 4 weeks prior to enrollment or anticipation that such a live attenuated vaccine will be required during the study
* Prior treatment with a cluster of differentiation (CD)137 agonists, anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA4), anti-programmed cell death 1 (PD-1), or anti-PD-L1 therapeutic antibody or pathway targeting agents
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin-2) within 4 weeks or five half-lives of the drug, whichever is shorter, prior to enrollment
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, anti-tumor necrosis factor agents) within 2 weeks prior to enrollment or anticipated requirement for systemic immunosuppressive medications during the trial

  * Patients who have received acute, low dose, systemic immunosuppressant medication (e.g., a one-time dose of dexamethasone for nausea) may be enrolled after a discussion and approval by the principal investigator
  * The use of inhaled corticosteroids and mineralocorticoids (eg, fludrocortisone) is allowed

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days after completion of study treatment
  Adverse events observed will be summarized in terms of type (organ affected or laboratory determination), severity (by National Cancer Institute CTCAE v4 and nadir or maximum values for the laboratory measures), time of onset (i.e. course number), duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects by dose and by course.
Response rate using irRECIST | Up to 30 days after completion of study treatment
  All responses will be reported. Response rate among patients with measurable disease will be summarized by exact binomial confidence intervals.
Progression free survival using RECIST 1.1 and irRECIST | From start of treatment to time of progression or death, whichever occurs first, assessed up to 30 days after completion of study treatment
  Progression free survival will be summarized with Kaplan-Meier plots to describe the outcome of patients treated on this protocol. The median progression free survival time will be estimated using standard life table methods.

OTHER OUTCOMES:
Changes in biomarkers | Baseline to up to 30 days after completion of study treatment
  Correlative biomarker endpoints (PD-L1, CD8, CD4, FoxP3) are exploratory and hypothesis generating. Descriptive statistics will be applied to characterize differences within a given patient pre-treatment to post-treatment and between responders and non-responders and to provide a preliminary estimate of prognostic value for survival and freedom from progression.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Kelly, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis, Sacramento, California, United States